CLINICAL TRIAL: NCT02057393
Title: Infrared Lymphangiography as a Method of Sentinel Node Identification
Acronym: SPY-SN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Colette Pameijer, Associate Professor of Surgery, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 247374
Record Dates: First submitted 2014-01-24; First posted 2014-02-07 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Melanoma; Sentinel Node
Keywords: Melanoma; Sentinel node biopsy; Indocyanine green; Real time lymphangiography
MeSH Terms: conditions — Melanoma | interventions — Indocyanine Green; Technetium-99; Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indocyanine Green (Experimental): Single arm study, each subject receives 0.9ml ICG, methylene blue and technetium 99.
  Interventions: Drug: Indocyanine green; Drug: Technetium99; Drug: Methylene blue

INTERVENTIONS:
Drug: Indocyanine green — Subjects receive 0.9ml of ICG subcutaneously about the primary melanoma. The ICG has an infrared signal that is detected with the SPY Elite system (Lifecell). The ICG travels through the lymphatics to the sentinel node.
  Other Names: IC-Green
Drug: Technetium99 — Technetium99 is a standard, widely used radiopharmaceutical that is injected subcutaneoulsy about the primary melanoma site. Lymphoscintigraphy is performed to identify the draining nodal basin, and a gamma probe is used in the operating room to track the radioactive signal and find the sentinel node.
  Other Names: Technetium99 sulfur colloid
Drug: Methylene blue — Subjects receive 0.5-2ml of methylene blue subcutaneously about the primary melanoma at the time of surgery. The sentinel node should turn blue, which is visible with the naked eye.

SUMMARY:
The initial treatment for most people with melanoma involves wide excision of the skin and sentinel node biopsy. As with other cancers, the status of the sentinel node provides important prognostic information to the patient and physician. Sentinel node biopsy was first developed using only a blue dye. Technetium99, a radioactive protein, was added later and provides the ability to image the patient and identify relevant lymph node basins. For the last 15 years or so, the standard method of SLN localization includes both tech99 and blue dye. While the rates of localization overall are excellent, these methods each have drawbacks. We are investigating a new method of finding sentinel nodes that uses a green dye that has an infrared signal. Our hypothesis is that indocyanine green (ICG) and real time lymphangiography is equivalent to technetium99 and methylene blue in identifying sentinel nodes (SLN) in patients with melanoma.

DETAILED DESCRIPTION:
Patients with melanoma of the trunk or extremities were prospectively enrolled in this trial. Patients with head and neck melanoma were excluded from this study based on our pilot experience. ICG is poorly visualized through muscle, and there seems to be high background uptake in the parotid gland; both of these features limit the utility of ICG and fluorescence imaging. All subjects had T1b or greater melanoma, and met current National Comprehensive Cancer Network (NCCN) guidelines for sentinel node biopsy. All subjects had injection of tech99 and lymphangiography prior to surgery, and injection of indocyanine green (ICG) and methylene blue dye (MB) in the operating room. We utilized methylene blue dye for all subjects due to poor availability of isosulfan blue for a period of time, and to maintain consistency in the trial. Up to 1ml of MB was injected, and 0.9ml ICG (2.5 mg/ml). The ICG and MB were injected into the dermis separately, after induction of anesthesia and prior to prepping the patient.

Each lymph node basin was examined with the gamma probe and imaged with the SPY Elite (Novadaq) prior to making skin incision, with assessment of the visibility of ICG through the skin (yes or no). Once incision was made, the basin was periodically imaged with SPY, or dissection was carried out with real time lymphangiography until the sentinel node was identified. The camera of the SPY machine is positioned over the basin, with the image projected onto a monitor. Similar to laparoscopy, the surgeon can watch the image and operate at the same time. Each sentinel node was assessed for the presence of each dye. A lymph node with any one of the dyes present was considered a sentinel node, and was resected. Fluorescence and blue dye were measured as yes or no, and not quantitated. Additional data collected includes demographic data, the dose of ICG and MB given, adverse effects from any dye, the total number of sentinel nodes identified and the number of malignant sentinel nodes. Pair-wise comparisons were made between the three dyes regarding the number of detected sentinel nodes, and the number of detected metastatic nodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed melanoma.
* All patients with melanoma of the arm, leg or trunk who qualify for a sentinel node biopsy based on the characteristics of their primary tumor are eligible to participate. Patients with melanoma that is T1b or greater are recommended to have a sentinel node biopsy.
* Age >18 years. Melanoma is extremely uncommon in children, this disease is not relevant in this age group.
* The effects of IC-Green on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with melanoma on the head or neck are excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IC-Green, sodium iodide or other agents used in the study.
* Pregnant women are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colette Pameijer, MD, Principal Investigator — Associate Professor of Surgery
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jain V, Phillips BT, Conkling N, Pameijer C. Sentinel lymph node detection using laser-assisted indocyanine green dye lymphangiography in patients with melanoma. Int J Surg Oncol. 2013;2013:904214. doi: 10.1155/2013/904214. Epub 2013 Dec 8. PMID 24382997

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indocyanine Green
Started | 89
Completed | 87
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Patient did not meet criteria | 1

BASELINE CHARACTERISTICS:
Population: 89 subjects were enrolled, one subject retracted consent, and another was deemed ineligible after enrollment, leaving 87 evaluable participants.
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 87
Age, Continuous [Median (Full Range); unit: years] | 65 [26 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87
BMI [Median (Full Range); unit: kg/m2] | 28 [17 to 51.5]

OUTCOME MEASURES:

1. Primary Outcome: Equivalence of ICG and Real Time Lymphangiography to technetium99 and Blue Dye in Localizing Sentinel Nodes
Description: The primary outcome measure is the accuracy of indocyanine green (ICG) and real time lymphangiography to identify sentinel nodes (SLN) in patients with melanoma, compared to tech99 and methylene blue. Tech99 is considered the standard, for comparison. Accuracy is being determined by the number of sentinel nodes that are identified with ICG, compared to tech99 or methylene blue.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: number of sentinel nodes per patient
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 87
number of sentinel nodes per patient | 1.87 (0.95)

ADVERSE EVENTS:
Time Frame: 2 weeks post-op
Arm/Group | Indocyanine Green
All-Cause Mortality (participants affected / at risk) | 0/87
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes